CLINICAL TRIAL: NCT01215409
Title: Vardenafil in Routine Treatment of Erectile Dysfunction
Brief Title: Real Life Safety and Efficacy of Vardenafil
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14328; LV0611TW (Other: Company internal)
Record Dates: First submitted 2010-09-28; First posted 2010-10-06 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Erectile Dysfunction
Keywords: Levitra; Erectile dysfunction; Taiwan
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — 5 mg or 10 mg or 20 mg of Vardenafil, orally when necessary for 2 months

SUMMARY:
In this uncontrolled, non-randomized, prospective, local post-marketed surveillance study, data are obtained on safety and efficacy of LEVITRA® in routine treatment of erectile dysfunction. The general objectives are to evaluate the product safety (primarily by recording adverse events), efficacy and patient acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient (>/=18 years) with erectile dysfunction treated with LEVITRA®.
* Patients must be able to give written informed consent for participation in the study after receiving detailed written and oral information prior to the study.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the product information (Package Insert).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
General assessment of patients concerning efficacy and tolerability of vardenafil treatment | 2 months

SECONDARY OUTCOMES:
Time to first intercourse after intake of vardenafil | 2 months
Percentage of successful second intercourse within 24 hours | 2 months
Percentage of participants who are willing to continue treatment | 2 months
Number of participants with adverse events | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Taiwan